CLINICAL TRIAL: NCT00577174
Title: Mitochondrial Function in Pediatric Obesity
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Lawson Wilkins Pediatric Endocrine Society (Other); Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Amy Fleischman, MD, Assistant Professor, Massachusetts General Hospital
Other Study IDs: 1K23DK080658 (NIH); 2006p001067, Partners IRB; 575, MIT IRB
Record Dates: First submitted 2007-12-18; First posted 2007-12-20 (Estimated); Last update posted 2012-04-30 (Estimated); Status verified 2012-04

CONDITIONS: Obesity; Insulin Resistance
Keywords: Children; Obesity; Insulin resistance; Diabetes; Mitochondrial Function
MeSH Terms: conditions — Obesity; Insulin Resistance; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Case-Control
Biospecimen Retention: Samples With DNA — Whole blood, serum, white blood cells
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1. Controls: Healthy children ages 8 to 18 years
- 2. Obese childrens: Obese children, ages 8 to 18 years

SUMMARY:
The prevalence of pediatric obesity is increasing at an unprecedented rate. Obese children are at risk for the development of insulin resistance, relative insulin deficiency and type 2 diabetes mellitus. However, the cause of insulin resistance remains an area of scientific interest. The study of type 2 diabetes in children is limited by the lack of a non-invasive method to evaluate insulin resistance. Recent studies have suggested that mitochondrial dysfunction is associated with, and perhaps predictive of insulin resistance in adult relatives of individuals with type 2 diabetes. Mitochondria generate energy in muscle tissue through the production of ATP, and are important in the metabolism of both glucose and fat. This study evaluates a novel, non invasive, safe method for predicting insulin resistance and diabetes in children using a magnetic resonance imaging (MRI) based technique to measure mitochondrial function. We propose to investigate mitochondrial function and glucose metabolism in obese and non-obese children in early, mid and late puberty. Analyses will be conducted to investigate the presence of mitochondrial dysfunction in obese children, to evaluate the contribution of mitochondrial dysfunction to insulin resistance, and to determine the contribution of pubertal status to mitochondrial dysfunction and insulin resistance. The successful completion of this study would provide evidence to support the hypothesis that mitochondrial dysfunction plays a role in insulin resistance and diabetes in children. In addition, it would provide a new technique for the prediction of disease states and perhaps lead to the development of preventative therapeutics for insulin resistance and type 2 diabetes in children.

We hypothesize that mitochondrial dysfunction will mirror the progression of insulin resistance and precede and predict abnormal glucose metabolism in a population with pediatric obesity

DETAILED DESCRIPTION:
Aim I: A cross sectional study to evaluate baseline mitochondrial function in obese children compared to non-obese children. Determine whether children with pediatric obesity have impaired mitochondrial function based on 31P magnetic resonance spectroscopy when compared to healthy non-obese control children.Examine the relationship between mitochondrial function and insulin resistance in obese and non-obese children. Determine the impact of pubertal stage on mitochondrial function in obese and non-obese children.

Aim II:A prospective evaluation to determine in a longitudinal cohort study the timing and relationship of mitochondrial dysfunction to the development of insulin resistance in prepubertal/early pubertal obese children compared to prepubertal/early pubertal non-obese children. Determine in a longitudinal cohort study if obese children with mitochondrial dysfunction develop greater insulin resistance and/or impaired glucose tolerance at an earlier time point. Evaluate the relationship of obesity, timing of puberty and related changes in hormone levels to mitochondrial function and the development of insulin resistance and/or impaired glucose tolerance in longitudinal analyses.

ELIGIBILITY:
Inclusion Criteria:

1. Girls and boys ages 8 to 18 years old
2. Non-obese cohort: body mass index less than 75th percentile for age
3. Obese cohort: body mass index more than 95th percentile for age

Exclusion Criteria:

1. Underlying medical problem with potential to affect growth, pubertal development or glucose homeostasis
2. Chronic medical therapy with glucocorticoids, growth hormone, estrogen, progesterone, testosterone, or other medications with the potential to alter growth, pubertal development or glucose homeostasis within the proceeding 6 months
3. Personal history of diabetes
4. Family history of diabetes in first degree relative
5. Inability to have MRI scan performed due to metal prosthesis or implant

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Healthy and obese children from clinical practices and the local community
Sampling Method: Non-Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2007-06; Primary Completion 2011-08 (Actual); Study Completion 2012-10 (Estimated)

PRIMARY OUTCOMES:
Determine whether children with pediatric obesity have impaired mitochondrial function based on 31P magnetic resonance spectroscopy when compared to healthy non-obese control children | 4 years
Examine the relationship between mitochondrial function and insulin resistance in obese and non-obese children | four years

SECONDARY OUTCOMES:
Determine the impact of pubertal stage, dietary intake, activity recall, inflammatory markers and metabolic markers on mitochondrial function in obese and non-obese children | four years
Evaluate the relationship of obesity, timing of puberty and related changes in hormone levels to mitochondrial function and the development of insulin resistance and/or impaired glucose tolerance in longitudinal analyses | four years

CONTACTS AND LOCATIONS:
Overall Officials: Amy D Fleischman, MD, MMSc, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Result] Fleischman A, Kron M, Systrom DM, Hrovat M, Grinspoon SK. Mitochondrial function and insulin resistance in overweight and normal-weight children. J Clin Endocrinol Metab. 2009 Dec;94(12):4923-30. doi: 10.1210/jc.2009-1590. Epub 2009 Oct 21. PMID 19846731
- [Result] Fleischman A, Makimura H, Stanley TL, McCarthy MA, Kron M, Sun N, Chuzi S, Hrovat MI, Systrom DM, Grinspoon SK. Skeletal muscle phosphocreatine recovery after submaximal exercise in children and young and middle-aged adults. J Clin Endocrinol Metab. 2010 Sep;95(9):E69-74. doi: 10.1210/jc.2010-0527. Epub 2010 Jun 16. PMID 20554709
- [Result] McCormack SE, McCarthy MA, Farilla L, Hrovat MI, Systrom DM, Grinspoon SK, Fleischman A. Skeletal muscle mitochondrial function is associated with longitudinal growth velocity in children and adolescents. J Clin Endocrinol Metab. 2011 Oct;96(10):E1612-8. doi: 10.1210/jc.2011-1218. Epub 2011 Aug 10. PMID 21832105